CLINICAL TRIAL: NCT01511432
Title: A Two-Part, Phase 1, Randomized, Open-Label, Crossover Study to Evaluate the Relative Bioavailability of 3 Novel Oral Formulations of Telaprevir Relative to Incivek 375-mg Tablets When Administered as a Single 1125-mg Dose to Healthy Subjects
Brief Title: A Study to Assess the Relative Bioavailability Three New Formulations of Telaprevir in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: VX11-950-025
Record Dates: First submitted 2012-01-09; First posted 2012-01-18 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Hepatitis C
Keywords: Relative bioavailability; telaprevir formulations
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Part A will be a 4-formulation, 4-sequence, 4-period crossover relative bioavailability study of 3 novel oral telaprevir formulations relative to the 375-mg Incivek tablet in the fed state.
  Interventions: Drug: telaprevir formulation A; Drug: telaprevir Formulation B; Drug: telaprevir Formulation C; Drug: telaprevir Formulation D
- Part B (Experimental): Part B will be a 2-formulation, 6-sequence, 3-period cross-over relative bioavailability study of the novel oral telaprevir formulation selected from Part A in the fasted relative to the fed state and relative to the 375-mg Incivek tablet in the fasted state
  Interventions: Drug: telaprevir formulation A; Drug: telaprevir Formulation B; Drug: telaprevir Formulation C; Drug: telaprevir Formulation D

INTERVENTIONS:
Drug: telaprevir formulation A — A single 1125-mg dose administered orally
Drug: telaprevir Formulation B — A single 1125-mg dose administered orally
Drug: telaprevir Formulation C — A single 1125-mg dose administered orally
Drug: telaprevir Formulation D — A single 1125-mg dose administered orally

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability, safety, and tolerability of 3 new formulations of telaprevir relative to the Incivek 375-mg tablets.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (male and female of non-childbearing potential) between the ages of 18 and 55 years
* Non-childbearing potential female subjects
* Male subjects and female partners must agree to use at least 2 methods of contraception
* Subjects with a body mass index (BMI) of 18 to 30 kg/m2 and weigh >50 kg at the Screening Visit.

Exclusion Criteria:

* Subjects with a positive test result for hepatitis B, hepatitis C, or HIV
* Subjects with a significant history of any illness, as deemed important by the investigator or any condition possibly affecting drug absorption
* Subjects with a positive urine screen for drugs of abuse
* Subjects with a history of regular alcohol consumption
* Subjects treated with an investigational drug within 30 days
* For Part A only: Subjects with 12-lead ECG QTcF >450 msec (males) or QTcF >470 msec (females) at the Screening Visit
* Subjects who use prescription and/or nonprescription medications or vitamins and/or dietary supplements
* Subjects who have made a blood donation of approximately 1 pint (500 mL) within 56 days prior to the first dose of study drug
* Subjects who have a female partner who is pregnant, nursing, or planning to become pregnant during the study or within 90 days of the last dose of study drug
* Subjects on hormone replacement therapy (HRT) must discontinue such therapy 28 days prior to the first dose of study drug
* Subjects who have a habit of using tobacco or nicotine containing products within 6 months before the Screening Visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
PK parameters: Maximum plasma concentration (Cmax), area under the concentration versus time curve (AUC) from time 0 to infinity (AUC0-∞) | Up to 57 days
• PK parameters: Maximum plasma concentration (Cmax), area under the concentration versus time curve AUC from time 0 to last time point (AUC0-tlast) | Up to 57 Days

SECONDARY OUTCOMES:
The safety and tolerability of 3 oral formulations of telaprevir as assessed by adverse events, serious adverse events and results of clinical laboratory tests (serum chemistry, hematology, and urinalysis), vital signs, and 12-lead electrocardiograms | Up to 57days
Time to reach Cmax after dosing (tmax) and terminal half-life (t1/2) of telaprevir | Up to 57 Days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Texas, Dallas, Texas
  - Wisconsin, Madison, Wisconsin